CLINICAL TRIAL: NCT04988451
Title: Family ASL: Longitudinal Study of Deaf Children and Hearing Parents Who Receive Services to Support the Learning of American Sign Language (ASL)
Brief Title: Family ASL: Longitudinal Study of Deaf Children and Hearing Parents Who Receive Services to Support the Learning of ASL
Acronym: FASL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Diane Lillo-Martin, BOT Distinguished Professor, University of Connecticut
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H20-0037; R01DC016901 (NIH)
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Deafness; Hearing Loss
Keywords: language; sign language; language development; child language; child, preschool; parents; caregivers
MeSH Terms: conditions — Deafness; Hearing Loss; Language; Sign Language

STUDY DESIGN:
Intervention Model Description: Single Case Design - interrupted time series. Participants will receive intervention in 6-week on/off blocks. Measurements are taken in both on and off weeks.
  The Bayesian procedure developed by Swaminathan et al. (2014) involves fitting piece-wise linear or curvilinear trends across the phases, modeling dependencies in the observations with a suitably chosen autoregressive error scheme, and using the Markov Chain Monte Carlo (MCMC) method to obtain the posterior distributions of the model parameters and effect size measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASL Services - Adult ASL Development (Experimental): Presence (or absence, across 6-week periods) of ASL services designed to support improvement in ASL fluency
  Interventions: Behavioral: ASL Services
- ASL Services - Child Language Development (Experimental): Presence (or absence, across 6-week periods) of ASL services designed to support improvement in ASL fluency
  Interventions: Behavioral: ASL Services

INTERVENTIONS:
Behavioral: ASL Services — ASL specialist meets with participants and provides ASL instruction

SUMMARY:
This study examines the development of American Sign Language by deaf and hard of hearing (DHH) children and their parents.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, adult participants who give written informed consent and children whose parents who give written permission will be enrolled in the study. They will participate in preliminary language tasks to assess baseline performance on American Sign Language (ASL) measures. Subsequently they will have weekly sessions with an ASL Specialist to support their development of ASL, following a 6-week on/6-week off ABABABAB sequence.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Children ages 2;00 - 2;11 at the start of the longitudinal project
* Child is Deaf/ Hard-of-Hearing
* Participating in a program utilizing a bimodal bilingual philosophy

Adults:

- One adult caregiver for each child

Exclusion Criteria:

* Children with previously-diagnosed conditions other than deafness known to affect language and cognitive development
* Families without access to internet (at home or other locations)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in ASL Phonological Production Accuracy over 12 Months | Baseline and 12 months
  Participants copy ASL signs produced on video; their productions are scored for phonological accuracy and reported as percent correct out of all possible phonological features. Weekly measures are taken for SCD analysis.

SECONDARY OUTCOMES:
Change from Baseline in ASL Production Frequency over 12 Months | Baseline and 12 months
  Participants engage in naturalistic play sessions which are videorecorded. Sessions are analyzed for the number of productions in ASL over a 15-minute period. Weekly measures are taken for SCD analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Diane C Lillo-Martin, Ph.D., Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut - Department of Linguistics, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from language tasks
Time Frame: After (or with) publication of the results
Access Criteria: De-identified numerical coding scores will be shared using an open science site that is generally accessible